CLINICAL TRIAL: NCT00038064
Title: A Randomized, Open-Label Study of Darbepoetin Alfa (Novel Erythropoiesis Stimulation Protein, NESP) and rHuEPO for the Treatment of Anemia in Subjects With Non-Myeloid Malignancies Receiving Multicycle Chemotherapy
Brief Title: Anemia in Patients With a Non-Myeloid Malignancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20010101; NCT00046982 (obsolete NCT alias)
Record Dates: First submitted 2002-05-28; First posted 2002-05-29 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Neoplasms; Anemia
Keywords: anemia of cancer/chemotherapy; non-myeloid malignancies; Drug Therapy
MeSH Terms: conditions — Neoplasms; Anemia | interventions — Darbepoetin alfa

ARMS (2):
- rHuEPO (Active Comparator)
  Interventions: Drug: rHuEPO
- Darbepoetin alfa (Experimental)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — Darbepoetin alfa will be administered 4.5 mcg/kg QW until hemoglobin correction is achieved. Subjects meeting hemoglobin criteria for correction will receive a maintenance dose of darbepoetin alfa of 4.5 mcg/kg Q3W.
  Arms: Darbepoetin alfa
Drug: rHuEPO — 150 IU/kg TIW
  Arms: rHuEPO

SUMMARY:
Chemotherapy can often cause anemia in patients with cancer. Anemia is a low number of red blood cells. The symptoms of anemia may include fatigue, dizziness, headache, chest pain, and shortness of breath. Erythropoietin is a hormone made by the kidneys that signals the bone marrow to produce more red blood cells. Recombinant human erythropoietin has been produced in the laboratory and has the same effect as the hormone produced by the body. Use of recombinant human erythropoietin allows the body to produce more red blood cells, possibly eliminating or decreasing your symptoms and the need for a red blood cell transfusion. Recombinant human erythropoietin is FDA approved to treat anemia in cancer patients receiving chemotherapy. This clinical study is investigating the effectiveness of darbepoetin alfa for the treatment of anemia in patients with non-myeloid malignancies who are receiving multicycle chemotherapy. Darbepoetin alfa is a recombinant erythropoietic protein that stimulates the production of red blood cells. This medication has not been approved to treat cancer patients with anemia, however it has been approved by the FDA to treat chronic renal failure patients with anemia.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of legal age, diagnosed with a non-myeloid malignancy and scheduled to receive at least 12 additional weeks of cyclic cytotoxic chemotherapy from the time of first dose of study drug
* Screening hemoglobin concentration less than or equal to 11.0 g/dL
* ECOG performance status of 0 to 2 (inclusive)

Exclusion Criteria:

* History of seizure disorder
* Primary hematologic disorder that could cause anemia
* Unstable or uncontrolled disease/condition related to or affecting cardiac function
* Clinical evidence of chronic infection/inflammatory disease
* Positive test for HIV infection
* Previously confirmed neutralizing antibodies to rHuEPO
* Received rHuEPO or darbepoetin alfa therapy within 4 weeks of study day 1 or more than 2 RBC transfusion occurences

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2002-01; Primary Completion 2003-10 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Time to first hemoglobin response during the treatment period | during the treatment period

SECONDARY OUTCOMES:
Overall incidence of adverse events, serious adverse events, and severe or life threatening adverse events | throughout study
Incidence, if any, of neutralizing antibody formation to study drug (darbepoetin alfa or rHuEPO) | throughout study
Average weekly dosage of study drug during the 16-week treatment period | 16-week treatment period
Receiving red blood cell (RBC) transfusion from week 5 to week 12 | from week 5 to week 12
Change in FACT-Fatigue scale score from baseline to week 7 | from baseline to week 7
Percentage of subjects who have a rapid rate of hemoglobin concentration rise and negative clinical consequences associated with this rise | throughout study
Profile of change in FACT-Fatigue scale score from baseline over the treatment period | from baseline over the treatment period
Change in FACT-Fatigue scale score from baseline to End of Treatment Period (EOTP) | from baseline to EOTP
Change in FACT-Physical Well-being scale score from baseline to EOTP | from baseline to EOTP
Receiving RBC transfusion during the treatment period | during the treatment period
Number of units of RBC transfused during the treatment period | during the treatment period
Achieving a hemoglobin response by week 7 | baseline to week 7
Change in hemoglobin concentration from baseline to EOTP | from baseline to EOTP
Time to first hematopoietic response | throughout study
Achieving a hemoglobin correction | throughout study
Number and percentage of subjects who exceed the hemoglobin concentration threshold | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20010101.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/